CLINICAL TRIAL: NCT07068438
Title: A Clinical Evaluation of the Pulsed Electric Field Ablation System for the Treatment of the Symptoms of Chronic Bronchitis in Adult Patients With COPD
Brief Title: Clinical Study of the Pulsed Electric Field Ablation System in Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hengruihongyuan Medical Technology Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COPD 1.0
Record Dates: First submitted 2025-06-23; First posted 2025-07-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chronic Bronchitis; COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Electric Field Ablation System (Experimental)
  Interventions: Device: Pulse electric field ablation system
- Sham Procedure (Sham Comparator)
  Interventions: Device: Sham Procedure

INTERVENTIONS:
Device: Pulse electric field ablation system — Bronchial rheoplasty (BR) is a staged procedure wherein pulsed electric fields are delivered to the right lung in the first treatment visit, and then the left lung is treated approximately 1 month later.
  Arms: Pulsed Electric Field Ablation System
Device: Sham Procedure — Staged sham procedure: the catheter is inserted into the right lung, but energy is not delivered; then the same steps are performed in the left lung approximately 1 month later (no energy is delivered to the patient).
  Arms: Sham Procedure

SUMMARY:
This is a prospective, randomized, parallel group, sham-controlled, multicenter clinical trial. The objective is to evaluate the safety and effectiveness of pulsed electric field ablation system manufactured by Suzhou Hengruihongyuan Medical Technology Co., Ltd. for the treatment of the symptoms of chronic bronchitis in adult COPD patients with moderate to severe chronic bronchitis. A total of 210 patients will be randomized into the experimental group and the sham group (2:1).

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age is ≥35 years and ≤80 years.
2. Patient has chronic bronchitis, defined as productive cough for three months in each of two successive years, whereas other causes of productive cough have been ruled out.
3. Patient has a CAT score ≥ 10.
4. Patient has an SGRQ score ≥ 25.
5. Patient's responses to the first two questions of the CAT instrument sum to ≥ 7 points or the sum is 6 points and the patient's total CAT score is > 20 points.
6. Patient has FEV1/FVC < 0.70.
7. Patient has a pre-procedure post-bronchodilator FEV1 percent predicted of ≥ 30%.
8. Patient is receiving guideline directed pharmacotherapy which includes one or more long acting bronchodilator (LAMA, LABA) with or without an inhaled corticosteroid for at least 8 weeks prior to randomization, unless the patient has attempted such therapy within the past 1 year without significant clinical response or had an adverse reaction.
9. In the opinion of the Primary investigator, patient is able to undergo 2 bronchoscopies under general anesthesia and is able to adhere to the study follow-up schedule.
10. Informed consent signed by the patient or legal representative.

Exclusion Criteria:

1. Patient has known unresolved lower respiratory tract infection (e.g., pneumonia, mycobacterium avium-intracellulare infection (MAI), fungus, tuberculosis).
2. Patient has a steroid-dependent condition requiring >10 mg of oral corticosteroid per day.
3. Patient has any implantable electronic device (e.g., pacemaker, cardioverter defibrillator) that cannot be turned off during the procedure.
4. Patient has a history of ventricular tachy-arrhythmia or clinically significant atrial tachyarrhythmia within the past two years, or sinus bradycardia with a heart rate of under than 45 beats per minute, unless the arrhythmia has been treated and/or patient is in regular rhythm during the screening phase.
5. Subject has lung cancer.
6. Patient has a pulmonary nodule or cavity that in the judgement of the Primary investigator may require intervention during the course of the study.
7. Patient had prior lung surgery, such as lung transplant, LVRS, lobectomy, lung implant/prosthesis, metal airway stent, valves, coils or bullectomy.
8. Patient has emphysema of greater than or equal to 50% as quantified on baseline HRCT scan as determined by the CT Core Lab.
9. Patient has asthma based on Global Initiative for Asthma (GINA) criteria.
10. Patient has clinically significant bronchiectasis influencing the patient's clinical symptoms of cough and phlegm.
11. Patient has actively smoked (including tobacco, marijuana, e-cigarettes, vaping, etc.) within the last 2 months.
12. Patient is unable to walk over 225 meters in 6 minutes.
13. Patient has a serious medical condition that, in the Primary investigator's opinion, could compromise patient safety or confound the interpretation of the patient's response to therapy (e.g., congestive heart failure, cardiomyopathy, or myocardial infarction in the past year, renal failure, liver disease, cerebrovascular accident within the past 6 months, uncontrolled diabetes (HbA1c >8%), uncontrolled hypertension (diastolic BP >100mmHg) or autoimmune disease requiring treatment with immunosuppressant medications or a disease requiring chemotherapy).
14. Patient has uncontrolled GERD.
15. Patient has known severe pulmonary hypertension (pulmonary artery SP ≥ 50 mmHg).
16. Patient has a known sensitivity to medication required to perform bronchoscopy (i.e., lidocaine, atropine, benzodiazepines).
17. Patient is pregnant, nursing, or planning to get pregnant during study duration.
18. Patient is currently participating in another clinical study involving an investigational product.
19. Patient is receiving anticoagulation for a cardiovascular indication and, in the Primary investigator's opinion, unable to suspend anticoagulant medications (i.e., aspirin, clopidogrel, warfarin) during bronchoscopy in accordance.
20. Patient has known airway colonization with drug-resistant bacteria such as Pseudomonas aeruginosa, methicillin-resistant Staphylococcus aureus, Burkholderia cepacia complex, Mycobacterium tuberculosis, Mycobacterium abscessus, Trichoderma, or other significant fungi.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) Score | 6 months
  Mean change from baseline in the COPD Assessment Test (CAT) total score, the total CAT score ranges from 0 to 40, where lower scores represent lower symptom burden

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) score | 3 and 12 months
  Mean change from baseline in the COPD Assessment Test (CAT) total score, the total CAT score ranges from 0 to 40, where lower scores represent lower symptom burden.
COPD Assessment Test (CAT) Score (items 1 and 2) | 3, 6 and 12 months
  Mean change from baseline in mean total scores for items 1 and 2 of the bilateral CAT scores (ranges from 0 to 10), where lower scores represent lower symptom burden.
St. George Respiratory Questionnaire (SGRQ-C) | 6 and 12 months
  Change from baseline in the total score of the COPD of the St. George Respiratory Questionnaire (SGRQ-C), the total score ranges from 0 to 100, where lower scores represent lower symptom burden.
Change from baseline in Modified Medical Research Council dyspnea scale (mMRC) scores | 3, 6 and 12 months
  Change from baseline in Modified Medical Research Council dyspnea scale (mMRC) scores, rated on a scale from 0 to 4, where lower grades represent lower symptom burden.
COPD Exacerbations | 12 months
  Rate of moderate and severe COPD exacerbations.
Pulmonary Function (FEV1) | 3, 6 and 12 months
  Changes from baseline in forced expiratory volume in the first second (FEV1) during a pulmonary function test (PFT).
Pulmonary Function (FEV1 /FVC ratio) | 3, 6 and 12 months
  Changes from baseline in the FEV1 /FVC ratio during a pulmonary function test (PFT).
The six minute walking test (6MWT) | 6 and 12 months
  Change from baseline in the 6-minute walk test.
Technical success rate | Approximately 15-minutes after device removal
  Success defined as:
  * Experimental group: Successful placement of the device, successful discharge, and successful withdrawal.
  * Control group: Successful placement of the device, and successful withdrawal.
  Calculation method: Patients with technical success/ total cases of subjects in the same group x 100%.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Anhui Chest Hospital, Hefei, Anui
  - Affiliated Beijing Chaoyang Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Hospital Emergency General, Beijing, Beijing Municipality
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second People's Hospital of Wuxi, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Sir Run Run Shaw Hospital, affiliated with Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang